CLINICAL TRIAL: NCT01890525
Title: PROMISE Substudy to Assess For Effective Dose of Radiation (PROMISE-SAFER), Specific Aim 3b
Brief Title: PROMISE Substudy to Assess For Effective Dose of Radiation (PROMISE-SAFER) Specific Aim 3b
Acronym: PROMISE-SAFER
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: R01HL109711-01 (NIH)
Record Dates: First submitted 2013-04-09; First posted 2013-07-01 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Chest Pain; Coronary Artery Disease; Angina
Keywords: radiation
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PROMISE study patients

SUMMARY:
The purpose of this study is to compare different methods of collecting the amount of radiation exposure patients receive in a clinical study. As part of the PROMISE study, the Duke Clinical Research Institute Outcomes and Follow-up Group will be contacting patients every six months to ask if they had any heart procedures or testing. This information will be used to estimate the amount of radiation that they may have received from heart testing being studied in this study, PROMISE-SAFER. Patients will be asked to collect information about each heart testing they receive during the time that they are enrolled in the PROMISE study. At the conclusion of the study, we will be able to determine which method was most accurate in collecting the amount of radiation exposure for this clinical study. Through this study we hope to develop an improved methodology to estimate cumulative radiation exposure from cardiac imaging. Comprehensive measurement of cumulative radiation exposure to patients may be critically important to minimize potential harm in future studies and in clinical practice.

ELIGIBILITY:
Inclusion Criteria: All patients who meet inclusion criteria and enroll in the parent PROMISE study will be eligible to participate in PROMISE-SAFER.

1. New or worsening chest pain syndrome or equivalent symptoms suspicious for clinically significant coronary artery disease
2. No prior evaluation for this episode of symptoms
3. Planned non-invasive testing for evaluation of possible coronary artery disease
4. Men age > 55 and women age ≥65 years
5. If age in men 45 - 54 or women 50 - 64 years, then must have increased probability of CAD due to EITHER:

   A. Diabetes Mellitus (DM) requiring medical treatment OR Peripheral Arterial Disease (PAD) defined as documented >50% peripheral arterial stenosis treated medically or invasively OR Cerebrovascular disease (stroke, documented > 50% carotid stenosis treated medically or invasively)

   OR

   B. At least one of the following cardiovascular risk factors:
   * Ongoing tobacco use
   * Hypertension
   * Abnormal ankle-brachial index defined as less than <0.9
   * Dyslipidemia
6. Serum creatinine < 1.5 mg/dL within the past 90 days
7. Negative urine/serum pregnancy test for female subjects of child-bearing potential and not breast-feeding

Exclusion Criteria:

1. Diagnosed or suspected acute coronary syndrome requiring hospitalization or urgent or emergent testing; Elevated troponin or creatinine kinase-MB
2. Hemodynamically or clinically unstable condition (systolic blood pressure < 90 mmHg, atrial or ventricular arrhythmias, or persistent resting chest pain felt to be ischemic despite adequate therapy)
3. Known coronary artery disease with prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass grafting or any angiographic evidence of coronary artery disease ≥50% lesion in a major epicardial vessel.
4. Any invasive coronary angiography or non-invasive anatomic or functional cardiovascular test for detection of coronary artery disease, including coronary computed tomographic angiography and exercise electrocardiogram, within the previous twelve (12) months.
5. Known significant congenital, valvular (> moderate) or cardiomyopathic process (hypertrophic cardiomyopathy or reduced systolic left ventricular function (left ventricular ejection fraction ≤ 40%)) which could explain cardiac symptoms.
6. Contraindication to undergoing a coronary computed tomographic angiography, including but not limited to:

   a. Pregnancy or breastfeeding
7. Life expectancy < 2 years
8. Unable to provide written informed consent or participate in long-term follow-up

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PROMISE study patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-08-01 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Methods to measure cumulative radiation exposure from a cardiac imaging trial will be compared to radiation measurements from the "gold standard" electronic medical records | 4 years
  In a single site (San Jose Medical Center - Kaiser Permanente) at a health maintenance organization where patients undergo all testing on site and comprehensive radiation records are maintained, 3 approaches to obtaining follow-up radiation dosimetry estimates will be compared: 1) the standard method used at all sites of combining those procedures identified on follow-up surveys with measured or imputed procedure dose estimates, 2) Radiation Log forms that patients will receive and will be asked to complete whenever they undergo further imaging, and 3) "gold standard" review of patient electronic medical records to identify all procedures with ionizing radiation and measured dose estimates from each procedure.

CONTACTS AND LOCATIONS:
Overall Officials: James J Jang, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- San Jose Medical Center - Kaiser Permanente, San Jose, California, United States